CLINICAL TRIAL: NCT02877186
Title: Effects of Non-nutritive Sweeteners on the Composition of the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Allison Sylvetsky (Meni), Assistant Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 011512
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Carbonated Water

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Diet Soda (Experimental): Consumption of diet soda three times daily for one week
  Interventions: Other: commercially-available diet soda
- Carbonated Water (Placebo Comparator): Consumption of plain, unsweetened, carbonated water three times daily for one week
  Interventions: Other: carbonated water (control)

INTERVENTIONS:
Other: commercially-available diet soda — Subjects are asked to consume diet soda three times daily for one week.
  Arms: Diet Soda
Other: carbonated water (control) — Subjects are asked to consume carbonated water three times daily for one week.
  Other Names: seltzer
  Arms: Carbonated Water

SUMMARY:
This pilot study is being conducted to evaluate whether consumption of diet soda sweetened with sucralose and acesulfame-potassium leads to changes in the gut microbiota. Following a one week run-in period, healthy, young adults are randomized to consume either diet soda or carbonated water (control) three times per day for one week. Stool and urine samples are collected at baseline, following the run-in, and after the one-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-35 years
* Consume less than 1 food/beverage with non-nutritive sweeteners per month
* Able and willing to consume diet soda three times daily for 1 week

Exclusion Criteria:

* Recent diet or significant weight change
* Antibiotic use in the past 3 months
* Diarrhea in the past two weeks
* Use of medications known to affect metabolism or weight
* Weight < 50 kg (110 lbs.)
* History of metabolic complications including high blood sugar, elevated cholesterol, or liver disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Taxa abundance before and after one-week of three times daily diet soda consumption | one week
  16S rRNA and metagenomics sequencing will be used to determine microbial composition of stool samples before and after the one week intervention.

REFERENCES:
- [Derived] Sylvetsky AC, Clement RA, Stearrett N, Issa NT, Dore FJ, Mazumder R, King CH, Hubal MJ, Walter PJ, Cai H, Sen S, Rother KI, Crandall KA. Consumption of sucralose- and acesulfame-potassium-containing diet soda alters the relative abundance of microbial taxa at the species level: findings of two pilot studies. Appl Physiol Nutr Metab. 2024 Jan 1;49(1):125-134. doi: 10.1139/apnm-2022-0471. Epub 2023 Oct 30. PMID 37902107
- [Derived] Sylvetsky AC, Walter PJ, Garraffo HM, Robien K, Rother KI. Widespread sucralose exposure in a randomized clinical trial in healthy young adults. Am J Clin Nutr. 2017 Apr;105(4):820-823. doi: 10.3945/ajcn.116.144402. Epub 2017 Feb 22. PMID 28228424